CLINICAL TRIAL: NCT02920528
Title: Subdissociative Dose Ketamine for Treatment of Acute Pain in Subjects With Chronic Pain: A Randomized Controlled Trial
Brief Title: Subdissociative Dose Ketamine for Treatment of Acute Pain in Subjects With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: United States Air Force Research Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Tanen, Professor of Emergency Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30612-01
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): placebo controlled arm
  Interventions: Drug: Placebo
- very low dose ketamine (Experimental): 0.25 mg/kg of sub-dissociative ketamine as an experimental arm
  Interventions: Drug: Ketamine
- low dose ketamine (Experimental): 0.50 mg/kg of sub-dissociative ketamine as an experimental arm
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — sub-dissociative ketamine
  Other Names: ketalar
  Arms: low dose ketamine; very low dose ketamine
Drug: Placebo — Normal Saline
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is a prospective, randomized controlled trial which will be conducted to determine whether sub-dissociative dose ketamine (SDDK) can improve pain control in subjects with chronic pain syndrome presenting to the emergency department with exacerbation of their chronic pain. The investigators also aim to determine whether use of SDDK can reduce the amount of subsequent opioid pain medications required for adequate pain relief in this population.

DETAILED DESCRIPTION:
1. The informed consent process will be initiated by investigators in the emergency department.
2. All potential subjects will be informed that participation in the study could lead to a positive urine drug test that could remain positive for up to a month after the conclusion of the study.
3. Female subjects of child bearing age, will have a pregnancy test performed prior to enrollment; any subjects who are pregnant will be excluded from this project.
4. Each subject will be asked to grade his/her pain severity on a 100mm non-hatched visual analog scale (VAS) ranging from 0 (no pain) to 100 (worst, maximum pain).
5. Each subject will be asked to fill out a baseline pain questionnaire
6. Each subject will be placed on monitors for continuous pulse oximetry, Heart Rate, Respiratory Rate, and blood pressure every 5 minutes for the duration of the study of one hour and longer for any patient who needs continued care. The patients temperature will be taken prior to the start of the protocol.
7. Each subject will have an intravenous catheter placed.
8. Each subject will be sequentially assigned to one of three treatment groups, based on a computer-generated randomization schedule, to receive an intravenous infusion of sub-dissociative Ketamine (0.25mg/kg), sub-dissociative dose Ketamine (0.5mg/kg), or an equal amount of normal saline.
9. All medications will be prepared by an emergency department pharmacist and all study medication intravenous bags will be identical in appearance and will be administered by the emergency department nurse caring for the patient who will be blinded to the study drug.
10. Each subject will receive lightly tinted sunglasses to wear during the duration of the study to minimize bias as ketamine can evoke a tell-tale short- lived nystagmus
11. Each subject will receive the study medication over a 20 minute period via an automated pump. At this point, the subjects will be asked to rate their pain on a VAS and asked if they need additional pain medication that will consist of intravenous hydromorphone with the dose and frequency determined by the discretion of the treating physician and documented on the data collection sheet.

ELIGIBILITY:
Inclusion Criteria:

* All adult subjects over the age of 18 with chronic pain* presenting to the emergency department with exacerbation of their chronic pain as their primary complaint
* Subjects who are willing and able to provide informed consent. *Chronic pain defined as greater > 3 months of symptoms and an initial VAS pain score > 70

Exclusion Criteria:

* History of overt psychosis, severe hypertension as defined by Systolic Blood Pressure > 180 mm Hg or Diastolic Blood Pressure >110 mm Hg, unstable angina, Coronary Artery Disease, Congestive Heart Failure, porphyrias, thyroid disease, seizure disorder, inability to provide informed consent: dementia, non-English/Spanish speakers, subjects in custody, suicidal, or clinically intoxicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tanen, MD, Principal Investigator — Los Angeles Biomedical Institute
Locations (1):
- Emergency Department, Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lumanauw DD, Youn S, Horeczko T, Yadav K, Tanen DA. Subdissociative-dose Ketamine Is Effective for Treating Acute Exacerbations of Chronic Pain. Acad Emerg Med. 2019 Sep;26(9):1044-1051. doi: 10.1111/acem.13755. Epub 2019 Apr 29. PMID 30901130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine
Started | 35 | 36 | 35
Completed | 32 | 35 | 30
Not Completed | 3 | 1 | 5
Not completed — Incomplete Data | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Did not meet inclusion criteria | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine | Total
Number analyzed (Participants) | 32 | 35 | 30 | 97
Age, Customized [Mean (Standard Deviation); unit: years] | 47.6 (15) | 44.3 (11.2) | 47.8 (11.5) | 46.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 18 | 57
  Male | 14 | 14 | 12 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 30 | 97
Baseline Pain as measured by validated Visualized Analog Scale (0 to 100 mm) [Mean (Standard Deviation); unit: units on a scale] | 91.2 (9.4) | 93.2 (8.9) | 91.4 (8.5) | 91.9 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Percentage of Subjects Who Achieved Significant Pain Relief Between the 3 Treatment Groups as Measured by a Visual Analog Pain Scale at 60 Minutes A Decrease of at Least 20 mm on the VAS Will be Considered "Significant" Pain Relief
Description: The primary endpoint was clinically significant pain relief defined a priori as a decrease in the pain VAS of at least 20 mm from baseline, which was arbitrarily chosen as the minimal amount that may be important to this group of patients and was extrapolated from studies of acute pain management in the ED. Using an effect size of 20-mm change in VAS as the marker for a successful outcome and the proportion of successes by group as the analysis point, we performed a power analysis using three groups: 0.5 mg/kg ketamine, 0.25 mg/kg ketamine, and placebo and found that a sample size of 96 subjects would be required to detect a statistically significant difference among groups with a power of 90% (a = 0.05). Expecting a loss of 10% of subjects due to patient withdrawal or incomplete data, 106 subjects were recruited. Only subjects who completed the 60-minute study and had data recorded for each of the time points were included in the analysis.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine
Number analyzed (Participants) | 32 | 35 | 30
Participants | 13 | 28 | 25

2. Secondary Outcome: Assess the Risk for Adverse Events Associated With Sub-dissociative Dose Ketamine
Description: Subjects will be continuously assessed for complications secondary to the sub-dissociative ketamine
Time Frame: 1 hour
Measure: Number; unit: recorded adverse events
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine
Number analyzed (Participants) | 32 | 35 | 30
recorded adverse events | 1 | 14 | 12

3. Post Hoc Outcome: Follow-up Pain Scores Obtained by Telephone at 24 - 48 Hours
Description: Subjects were contacted by phone 24 - 48 hours after the completion of the study infusion. Subjects were asked to score their pain on 10-point numeric rating scale where 0 represented no pain and 10 represented the worst pain they could be having. Pain score was recorded in increments of 1 from 0 - 10. Results were compared between groups using the Mann-Whitney U-test.
Time Frame: 24 - 48 hours after study drug infusion
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine
Number analyzed (Participants) | 30 | 31 | 28
units on a scale | 5 [4 to 8] | 5 [4 to 7] | 6 [3 to 8]

ADVERSE EVENTS:
Time Frame: Up to 48 hours after study enrollment
Arm/Group | Placebo | Very Low Dose Ketamine | Low Dose Ketamine
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/35 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/32 | 14/35 | 12/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Very Low Dose Ketamine (N=35) | Low Dose Ketamine (N=30)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) — Patients self-reported feeling nauseated
Dizziness (Nervous system disorders) | 1 (1) | 8 (8) | 3 (3) — Subjects were asked if they felt "dizzy"
Hallucinations (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) — Subjects were assessed for hallucinations
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety and Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Anxiety and Palpitations (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphoria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT02920528/Prot_SAP_000.pdf